CLINICAL TRIAL: NCT02166684
Title: The Potential of Do-it-yourself Devices for Obtaining Personal Health Data - P4@TNO Pilot Study
Brief Title: The Potential of Do-it-yourself Devices for Obtaining Personal Health Data
Acronym: P4@TNO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: W.J. Pasman (Other)
Responsible Party: Sponsor-Investigator, W.J. Pasman, PhD, TNO
Organization: TNO (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: P9608
Record Dates: First submitted 2014-06-16; First posted 2014-06-18 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Self-monitoring of Health; Health Behaviour Change
Keywords: Do-it-yourself devices; User-experiences; Health behavior; Self-measurement; Methodology, Evaluation; Personal health records; Blood Glucose Self-Monitoring; Self Blood Pressure Monitoring
MeSH Terms: conditions — Health Behavior | interventions — Blood Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Do-it-yourself devices (Experimental): All subjects will use do-it-yourself devices for self-monitoring health parameters
  Interventions: Device: Do-it-yourself devices

INTERVENTIONS:
Device: Do-it-yourself devices — Medisana Vifit is worn every day all-day by each subject
  Subjects use Medisana MTX Blood pressure monitor twice per week for 13 weeks to measure their blood pressure.
  Blood cholesterol is measured by subjects using the Mission Cholesterol 3-1 meter once at baseline and once after 13 weeks
  Subjects use Medisana BS 440 BT scale daily
  In three weeks (week 1, week 7 and week 13) subjects self-record food intake at three days (two week days and on weekend day) using the FatSecret app.
  Subjects self-measure fasting blood glucose twice per week for 13 weeks.
  Subjects perform a do-it-yourself Oral Glucose Tolerance Test in week 1 and week 13. Subjects use the Medisana MediTouch 2 for assessing blood glucose levels at t=0, t=30, t=60, t=90 and t=120.
  Other Names: Medisana Vifit - advanced activity tracker; Medisana MTX Blood pressure monitor - systolic and diastolic blood pressure; Medisana BS 440 BT scale - body weight; Medisana MediTouch 2 - blood glucose meter; FatSecret app - food intake application; Mission Cholesterol 3-1 meter - blood cholesterol level; Do-it-yourself Oral Glucose Tolerance Test

SUMMARY:
The study aims to evaluate whether do-it-yourself devices for self-measuring health parameters by subjects can be used for obtaining useful data in scientific studies.

Besides, the study aims to evaluate if increased awareness of own health status by self-monitoring health parameters also serves as motivational instrument for changing health behaviour.

DETAILED DESCRIPTION:
During this three month study subjects will self-monitor multiple parameters of health with do-it-yourself devices. Subjects are supplied with devices for measuring physical activity, food intake, body weight, blood pressure, blood glucose level and blood cholesterol level. These devices have to be used with varying frequencies, ranging from continuously to only a baseline- and endpoint measure.

Subjects will have to upload data resulting from these self-measures to an encoded account on an online portal.

At any time during the study, subjects can log-on to this portal, to gain insight in their own health parameters.

Only encoded subject data can be exported from this portal for data analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Age ranging from 18 - 67 years
2. Desk-job and not exceed the Dutch Standard of Healthy Physical Activity of 5 hours/week
3. Healthy as assessed by the Health and Lifestyle questionnaire
4. Body mass index: 20 - 30 kg/m2
5. Able to use self-monitoring devices
6. Voluntary participation
7. Having given written informed consent
8. Willing to comply with study procedures
9. Willingness to share pseudonymised data on food intake with external party Fatsecret (food intake app provider)
10. Willingness to share pseudonymised data on blood glucose, blood pressure, physical activity and body weight with external party Medisana (provider of measurement Toolkit)
11. Willingness to share pseudonymised data on food intake, blood glucose, blood cholesterol, blood pressure, physical activity and body weight with the Nutrition Research Cohort (NRC) database
12. Willing to accept use of all nameless data, including publication, and the confidential use and storage of all data by TNO
13. Have a desktop or laptop with internet access at home
14. Subjects should own a Smartphone with Bluetooth that runs either a recent version of iOS or Android.
15. Having one of the TNO locations in Delft, Den Haag or Rijswijk as posting

Exclusion Criteria:

1. Use of concomitant medication including medication known for its effects on blood glucose, cholesterol or insulin
2. Having a history of medical or surgical events that may significantly affect the study outcome, including physical limitations or cardio-vascular events
3. Having a pacemaker
4. Currently suffering from diabetes type I or type II as determined by the general practitioner
5. Reported slimming or medically prescribed diet
6. Physical, mental or practical limitations in using computerized systems
7. Alcohol consumption > 28 units/week for males and > 21 units (drinks)/week for females
8. Reported unexplained weight loss or gain of > 2 kg in the three months prior to the pre-study screening
9. Partner or first or second-degree relative from TNO personnel stationed at a TNO location in Zeist, Leiden, Hoofddorp or Soesterberg where the study protocol was developed.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Percentage of complete datasets | end of study (after 13 weeks)
  percentage is calculated for total complete datasets as well as complete datasets per device
Health behaviour change | baseline and after 13 weeks (end of study)
  established by comparing baseline values for food intake and physical activity as measured by a Lifestyle-questionnaire
User-experiences with do-it-yourself devices | after 13 weeks (end of study)
  as measured by a questionnaire on user-experiences as well as focus group interviews for more in-depth information

SECONDARY OUTCOMES:
self-measured blood pressure | baseline + weekly from week 1 until week 13
self-recorded food intake | week 1, week 7 and week 13
  every of the three periods, food intake will be recorded at two week days and one weekend day
daily physical activity | daily during 13 weeks (baseline - end of study)
  wearable activity tracker that measures number of steps taken, duration of activity and estimates the number of calories burned
Fasting blood glucose level | twice per week at baseline and from week 1 until 13
  self-assessed after overnight fast (at least eight hours)
body weight | three times per week at baseline and from week 1 to 13
  self-assessed with a smart scale that also calculates BMI and body fat percentage
blood cholesterol levels | baseline and after 13 weeks (end of study)
  self-assessed
oral glucose tolerance test (OGTT) | week 1 and week 13
  do-it-yourself version of OGTT; blood glucose levels will be assessed using the Medisana MediTouch 2
change in vitality as assessed with a vitality questionnaire (Vita-16) | baseline and week 13
change in subjective stress level as assessed with DASS-21 questionnaire | baseline and week 13
change in subjective quality of life as assessed with RAND-36 questionnaire | baseline and week 13

CONTACTS AND LOCATIONS:
Overall Officials: Wilrike J Pasman, PhD, Principal Investigator — Netherlands Organisation for Applied Scientific Research (TNO); Ben van Ommen, Dr. ir., Study Director — Netherlands Organisation for Applied Scientific Research (TNO)
Locations (1):
- Netherlands Organisation for Applied Scientific Research (TNO), Zeist, Utrecht, Netherlands